CLINICAL TRIAL: NCT05729711
Title: TEZSPIRE Subcutaneous Injection 210mg Specific Use-results Study (Long Term) in Patients With Bronchial Asthma.
Brief Title: TEZSPIRE (Tezepelumab) Asthma Japan Post-Marketing Study (PMS)
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5180C00034
Record Dates: First submitted 2023-02-07; First posted 2023-02-15 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Bronchial Asthma (Only the Patients With Severe or Intractable Bronchial Asthma Which Could Not be Controlled With the Existing Therapy)
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

SUMMARY:
The purpose of the investigation is to confirm the followings under the post-marketing actual long-term use of Tezspire.

1. Development of related AEs
2. Contributing factors possibly having an impact on the safety and effectiveness
3. Development of unexpected related AEs

DETAILED DESCRIPTION:
The purpose of the investigation is to confirm the followings under the post-marketing actual long-term use of Tezspire.

1. Development of related AEs
2. Contributing factors possibly having an impact on the safety and effectiveness
3. Development of unexpected related AEs

This investigation will be conducted to support the application for re-examination specified in Article 14-4 of the Act on Securing Quality, Effectiveness and Safety of Products Including Pharmaceuticals and Medical Devices.

ELIGIBILITY:
Inclusion Criteria:

* The evaluable patients are those treated with Tezspire for the first time due to "Bronchial asthma (only the patients with severe or intractable bronchial asthma which could not be controlled with the existing therapy)

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The evaluable patients are those treated with Tezspire for the first time due to "Bronchial asthma (only the patients with severe or intractable bronchial asthma which could not be controlled with the existing therapy)
Sampling Method: Non-Probability Sample
Enrollment: 416 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2029-11-16 (Estimated); Study Completion 2029-11-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of ADRs | 156 weeks
  the incidence of ADRs related to Tezspire Safety Specifications: Serious hypersensitivity, infection, malignancy, cardiac disorders

CONTACTS AND LOCATIONS:
Overall Officials: Toshimitsu Tokimoto, Study Director — AstraZeneca KK
Locations (34):
- Japan (34):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kagawa
  - Research Site, Kanagawa
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Nara
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saitama
  - Research Site, Shimane
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokyo
  - Research Site, Toyama
  - Research Site, Wakayama
  - Research Site, Yamagata
  - Research Site, Yamaguchi
  - Research Site, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA P harma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home